CLINICAL TRIAL: NCT03038802
Title: A Randomised Controlled Phase 1 Study of Vaccine Therapy for Control or Cure of Chronic Hepatitis B Virus Infection
Acronym: HBV003
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vaxine Pty Ltd (Industry)
Collaborators: Australian Respiratory and Sleep Medicine Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HBV003
Record Dates: First submitted 2017-01-30; First posted 2017-02-01 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Engerix-B

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, the investigator and outcomes assessors will be blinded as to which vaccine the subject has received
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard vaccine (Active Comparator): Subjects will receive regular intramuscular injections of a commercial hepatitis B vaccine (HBsAg containing aluminium hydroxide adjuvant) according to the same study schedule as the subjects in the experimental arm
  Interventions: Biological: Commercial Hepatitis B vaccine
- Experimental therapeutic vaccine (Experimental): Subjects will receive regular intramuscular injections of the experimental therapeutic hepatitis B vaccine (preS HBsAg containing Advax-2 adjuvant) in two cycles with the first cycle of four immunisations administered on days 0, 14, 28, 42. and the second cycle of four immunisations on days 70, 84, 98, and 112.
  Interventions: Biological: Therapeutic hepatitis B vaccine

INTERVENTIONS:
Biological: Therapeutic hepatitis B vaccine — HBV vaccine based on unique combination of recombinant PreS hepatitis B surface antigen particles formulated with Advax-2 adjuvant
  Other Names: Hepadvax(TM)
  Arms: Experimental therapeutic vaccine
Biological: Commercial Hepatitis B vaccine — Commercially available prophylactic hepatitis B vaccine formulated with alum adjuvant
  Other Names: Engerix B
  Arms: Standard vaccine

SUMMARY:
This is a pilot study to determine the safety and efficacy of a novel adjuvanted hepatitis B virus (HBV) vaccine formulated as a potential therapeutic vaccine against chronic HBV infection. An ongoing human clinical trial of this HBV vaccine in a prophylactic setting has confirmed this vaccine to be more effective at inducing seroconversion as measured by development of Hepatitis B surface antibody (HBsAb) in poor responder subjects than the standard alum-adjuvanted HBV vaccine, providing promise that this new vaccine may also be able to induce HBV viral control and/or seroconversion in chronically infected subjects

DETAILED DESCRIPTION:
Prophylactic immunisation with HBsAg-based vaccines leads to development of HBsAg antibodies that provide protection against HBV infection. Modern HBV vaccines are based on recombinant HBsAg produced by expression in yeast expression systems. For infants whose mothers are HBsAg positive, the first HBV vaccine dose is given at birth and three further doses are administrated during the following 12 months at 2, 4 and 6 or 12 months. Studies have shown that these HBV vaccines are 90 to 95% effective in preventing children from developing chronic infection if they have not yet been infected. Since 1982 over one billion doses of HBV vaccine have been used worldwide. However a number of groups have poor responses to the existing HBV vaccines and these include older adults (age > 40) and patients with immunodeficiency, diabetes or renal impairment. A pilot clinical study demonstrated that standard anti-HBV vaccination could reduce HBV replication in 50% of chronic carriers. A multicentre trial, showed both the efficacy and the limitations of this approach. This study included 118 treatment-naive patients, with detectable serum HBV DNA using a standard liquid hybridization study and biopsy-proven chronic hepatitis pre-vaccination. Over a 12-month period, they were given either five intradermal injections of 20 µg of a pre S2:S HBV vaccine (GenHevac B.Pasteur-Merieux) or a standard HBV vaccine (Recombivax, MSD) or no treatment. Three months after the first three vaccine injections, the percentage of serum HBV DNA negativity was higher in the vaccine groups (15.5%) than in the control group (2.7%). After 1 year follow-up and five vaccine injections, there was no difference in the rate of serum HBV DNA negativity, but those receiving HBV vaccines had significantly decreased HBV viral load between 6 and 12 months when compared to the control group. The rate of HBe:anti-HBe seroconversion did not differ between the vaccinated and unvaccinated groups, but early HBeAg negativity and anti-HBe detection after 6 months of follow-up was seen only in vaccinated patients (8 and 15% in groups B (Recombivax.) and C (GenHevac B.), respectively, compared with 0% in the controls). Analysis of the vaccine-induced immune responses in 40 patients with HBV chronic hepatitis during this vaccine trial showed that vaccination elicited T cell proliferative responses in 7 of 27 patients who received the vaccine versus none of the unvaccinated control group. These specific responses for envelope antigen were mediated by CD4 T cells that produced high levels of gamma interferon. The reduction of serum HBV-DNA in some of these patients suggests that induction of CD4 T cell responses could be important in controlling viremia after vaccine therapy of HBV chronic carriers.

Experiments in transgenic mice that constitutively express HBV in the liver as a model of asymptomatic chronic HBV carriers have shown that immunization can overcome functional tolerance to HBV by inducing a specific antiviral immune response. The study vaccine was tested for its ability to induce seroconversion in a HBV transgenic mouse model. The results confirmed that the vaccine induced a high titre of anti-HBsAg antibodies and suppressed HBV virus load in the liver. Importantly from a safety perspective no evidence of a flare in liver disease as reflected by elevation of liver functions tests, was seen despite evidence the vaccine suppressed liver virus. The vaccinated mice had the lowest levels of liver transaminases, consistent with the vaccine reducing virus-mediated damage to the liver.

This study will test the hypothesis that the investigational vaccine will boost HBV antibody and T cell responses in chronically infected patients and thereby improve HBV viral control and opportunity for seroconversion. As this is an exploratory study, subjects with chronic HBV infection will be enrolled whether or not they are on current antiviral treatment. This will then allow comparison of vaccine effects in subjects on and off concomitant antiviral treatment, with this data used to assist the design of future studies. The study will test the hypothesis that a potent preS HBV vaccine including Advax adjuvant will enhance both humoral and cellular immunity thereby helping to control chronic hepatitis B infection. The ultimate goal is to induce HBsAg seroconversion and effect permanent clearance of HBV or at a minimum to enable better immune control of viral replication. This pilot study will collect preliminary data on the safety and efficacy of this vaccine approach in chronically HBV infected individuals, as a precursor to larger efficacy studies in the future.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years of age or older
* Current evidence of HBV chronic infection (with or without cirrhosis) as indicated by detection of HBsAg and/or Hepatitis B DNA (Subjects on current nucleoside therapy may have no detectable Hep B DNA)
* If child bearing age, using contraception (barrier method, IUD or oral contraception)
* Able to provide written informed consent
* Willing and able to comply with the protocol for the duration of the study.

Exclusion Criteria:

* Positive for antibody to hepatitis B core antigen (anti-HBc) IgM with negative results for the rest of the HBV markers, indicating acute infection,
* Positive for anti-delta virus, or anti-hepatitis C virus or HIV
* Childs Pugh Score for Cirrhosis Mortality of Child grade B or greater
* Liver transaminases greater than 5 times the upper limit of normal
* History of severe allergic reaction to hepatitis B vaccine.
* Pregnancy or female of child-bearing age not using effective method of contraception.
* Presence of any other organ-specific disease that in the opinion of the investigator may result in risk to the subject from involvement in the study
* Current alcohol or drug abuse that in the opinion of the investigator may result in non-compliance.
* Participation in another clinical trial with an investigational agent within 30 days preceding initiation of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety assessment: Frequency of vaccine-related adverse events relative to active comparator vaccine | 12 months post immunisation
  Frequency of vaccine-related adverse events relative to active comparator vaccine
Viral load | 1 and 12 months post final immunisation
  Suppression of HBV viral load

SECONDARY OUTCOMES:
Seroconversion | 1 and 12 months post final immunisation
  Seroconversion to e antigen (if anti HBe negative at baseline) and seroconversion to surface antigen
T-cell response | 1 and 12 months post final immunisation
  Development of memory T-cell responses to HBV
B cell response | 1 and 12 months post final immunisation
  Development of memory B-cell responses to HBV

CONTACTS AND LOCATIONS:
Overall Officials: Nikolai Petrovsky, MBBS/PhD, Study Director — Vaxine Pty Ltd
Locations (1):
- ARASMI, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Undecided